CLINICAL TRIAL: NCT01539889
Title: Phase-I Study of Radiolabeled DFH-12 (PulmoBind) for Molecular Imaging of the Pulmonary Circulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: The PulmoBind Safety Trial
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease; Pulmonary Hypertension
MeSH Terms: conditions — Lung Diseases; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DFH-12 PulmoBind (Experimental): DFH-12 PulmoBind - 3 doses of; 5mCi for 5 subjects, 10mCifor 5 subjects and 15mCi for 10 subject
  Interventions: Radiation: 99mTC-PulmoBind

INTERVENTIONS:
Radiation: 99mTC-PulmoBind — DFH-12 (PulmoBind) is a peptide derived from human adrenomedullin (hAMI-52). Adrenomedullin (AM) is a 52-amino acid peptide produced by many tissues in the body, including the vascular endothelium. 3 radiolabeled doses of PulmoBind will be used in this study (5mCi, 10mCi and 15mCi) 5 healthy subjects per dose for the 5 mci and the 10 mci groups but 10 subjects will be used for the 15 mci group.

SUMMARY:
Pulmonary hypertension (PH) can be the result of various clinical conditions. It may be idiopathic or associated with various cardiovascular and lung disorders. Currently there is no test that can non-invasively detect abnormalities of the pulmonary circulation. There is a growing need for a non-invasive method to detect PH. There currently exists only ne agent approved in Canada for clinical imaging of the pulmonary circulation, 99mTc-labeled macroaggregates. This agent is exclusively used for the diagnosis of physical defects of the circulation due to pulmonary embolus. This agent is larger than small pulmonary vessels, limiting its sensitivity to detect small vascular defects, as well as potential infectious risks since albumin macroaggregates are derived from human albumin. There is need then for new lung tracers that could provide a greater safety profile while enabling functional as well as anatomical imaging of the pulmonary circulation. DFH-12 (PulmoBind) is a peptide derived from human adrenomedullin (hAMI-52). Hence the development of this novel AM derivative, PulmoBind, for molecular imaging of the pulmonary circulation. PulmoBind is labeled with 99mTc, the most commonly used imaging isotope in nuclear medicine.

ELIGIBILITY:
Inclusion Criteria:

* male or female greater than 18 years of age. Female subjects must be post-menopausal (defined as two years after menstrual cycle)
* within normal range for the following: BP systolic 100-140 mmHg and diastolic 50-90 mmHg;
* HR 60-100 beats per minute;
* oral temperature less than 37.6 degrees Centigrade;
* respiratory rate 12-20 breaths per minute;
* normal lung function tests;
* normal echocardiogram including estimation of pulmonary artery systolic pressure;
* normal chest x-ray; Normal electrocardiogram

Exclusion Criteria:

* any known chronic or acute medical condition with or without the need for chronic pharmacologic therapy or any condition that may interfere with normal biodistribution of DFH-12. Includes but not limited to:

  * lung parenchymal or lung vascular diseases such as chronic obstructive pulmonary disease,
  * bronchitis,
  * lung cancer,
  * pleural effusion,
  * emphysema,
  * asthma,
  * pulmonary fibrosis,
  * occupational lung disease,
  * pulmonary hypertension (primary or secondary),
  * systemic hypertension,
  * diabetes,
  * cancer,
  * kidney disease,
  * liver disease,
  * heart failure or previous myocardial infarction,
  * coronary artery disease,
  * peripheral vascular disease or inflammatory disease;
* subjects requiring chronic administration of any substance for a medical condition, active smoking or history of smoking for more than one year in the past 10 years, known self-reported alcoholism (active or abstinent);
* unable to tolerate study procedures ex.(venipuncture, movement restrictions during imaging);
* previous nuclear study since one week (to avoid cross-contamination)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To determine optimal dose of PulmoBind to be administered for lung imaging in humans | 48 hours
  To determine the optimal dose of Pulmobind by evaluating the safety and efficacy in three groups of subjects with 3 different doses of study drug; 5mCi, 10mCi, and 15 mCi.For safety evaluation we will provide pharmacokinetic and biodistribution data following injections of the 3 doses mentioned. Vital signs, hematology and biochemistry will also be captured for each of the doses up to 24 and 48 hours after injections of PulmoBind. Furthermore local and systemic reactions 24 hours and 48 hours after injections of PulmoBind will also be captured.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Dupuis, MD, Study Director — Montreal Heart
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Levac X, Harel F, Finnerty V, Nguyen QT, Letourneau M, Marcil S, Fournier A, Dupuis J. Evaluation of pulmonary perfusion by SPECT imaging using an endothelial cell tracer in supine humans and dogs. EJNMMI Res. 2016 Dec;6(1):43. doi: 10.1186/s13550-016-0198-3. Epub 2016 May 27. PMID 27234509
- [Derived] Harel F, Levac X, Nguyen QT, Letourneau M, Marcil S, Finnerty V, Cossette M, Fournier A, Dupuis J. Molecular imaging of the human pulmonary vascular endothelium using an adrenomedullin receptor ligand. Mol Imaging. 2015;14. doi: 10.2310/7290.2015.00003. PMID 25812438